CLINICAL TRIAL: NCT01624974
Title: A Double-Blind, Randomized, Placebo-Controlled, Multicenter, Crossover Study of MK-1029 in Adult Subjects With Persistent Asthma Who Remain Uncontrolled While Being Maintained on Montelukast
Brief Title: Study to Evaluate the Effectiveness and Safety of MK-1029 in the Treatment of Persistent Asthma That is Not Controlled With Montelukast (ML) in Adults (MK-1029-011)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1029-011; 2012-000642-35 (EudraCT Number); MK-1029-011 (Other: Merck Protocol Number)
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Results first posted 2018-11-23 (Actual); Last update posted 2019-01-02 (Actual); Status verified 2018-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — montelukast

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- MK-1029/Placebo (Experimental): Participants received 4 weeks treatment with MK-1029 150 mg once daily (QD) + ML 10 mg QD in Period III and Placebo QD + ML 10 mg QD in Period V. Period IV was a 4-week wash-out period during which participants received single-blind Placebo QD and open-label ML 10 mg QD.
  Interventions: Drug: MK-1029; Drug: Placebo; Drug: Montelukast (ML)
- Placebo/MK-1029 (Experimental): Participants received 4 weeks treatment with Placebo QD + ML 10 mg QD in Period III and MK-1029 150 mg QD + ML 10 mg QD in Period V. Period IV was a 4-week wash-out period during which participants received single-blind Placebo QD and open-label ML 10 mg QD.
  Interventions: Drug: MK-1029; Drug: Placebo; Drug: Montelukast (ML)

INTERVENTIONS:
Drug: MK-1029 — MK-1029 150 mg tablets taken QD
Drug: Placebo — Placebo tablets (matching the MK-1029 150 mg tablets) QD
Drug: Montelukast (ML) — ML 10 mg tablets QD

SUMMARY:
The purpose of this study is to evaluate the effect of MK-1029 on lung function in the treatment of adults who have persistent asthma that is uncontrolled with the use of montelukast (ML). Participants will use randomized study drug (either MK-1029 or placebo) for two separate 4-week treatment periods. All participants will also use ML during the treatment periods. The primary hypothesis is that MK-1029 is superior to placebo in change from baseline in forced expiratory volume in one second (FEV1) at the end of the 4-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* not pregnant or breastfeeding and does not plan to become pregnant for the duration of the study;
* symptoms of persistent asthma for at least one year;
* current use of asthma treatments: 1) "as-needed" inhaled SABAs (albuterol/salbutamol) and no asthma controller for at least 4 weeks prior to Screening Visit OR 2) stable dose of ICS, combination ICS/LABA and/or oral asthma controller(s) for at least 4 weeks prior to Screening Visit and able to tolerate discontinuing all controllers while receiving ML;
* no history of smoking OR no smoking for at least 1 year, with a smoking history of no more than 10 pack-years;
* able to maintain a constant day/night, awake/sleep cycle;
* agrees to not change habitual consumption of beverages or foods containing caffeine throughout the study;
* Body Mass Index (BMI) of 15 kg/m^2 to 40 kg/m^2.

Exclusion Criteria:

* history of myocardial infarction, congestive heart failure, or uncontrolled cardiac arrhythmia within 3 months prior to Screening Visit;
* hospitalized or hospitalization within 4 weeks prior to Screening Visit;
* intention of moving or anticipation of missing any study visits;
* any major surgical procedure(s) within 4 weeks prior to Screening Visit;
* participation in a clinical trial involving an investigational drug within 4 weeks prior to Screening Visit;
* current regular use or a recent past abuse (within past 5 years) of alcohol (>14 drinks/week) or illicit drugs;
* donation of a unit of blood within 2 weeks prior to Screening Visit or intention of donating a unit of blood during the study;
* evidence of another active pulmonary disorder such as bronchiectasis or COPD;
* treatment in an emergency room for asthma within 4 weeks prior to Screening Visit or hospitalization for asthma within 2 months prior to Screening Visit;
* respiratory tract infection which required treatment with antibiotics within 2 months prior to Screening Visit;
* evidence of active sinus disease within 1 week prior to Screening Visit;
* history of a psychiatric disorder, other than stable depression, within 3 months prior to Screening Visit;
* history of human immunodeficiency virus (HIV);
* hypersensitivity or intolerance to inhaled beta-agonists and/or leukotriene inhibitors or any of their ingredients, including lactose and galactose;
* unstable disease of the ophthalmologic, neurological, hepatic, renal, connective tissue, genitourinary, gastrointestinal, cardiovascular or hematologic systems;
* cancer (except for successfully treated basal and squamous cell carcinomas of the skin) or history of cancer within 5 years prior to Screening Visit;
* uncontrolled hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2012-08-09 (Actual); Primary Completion 2014-05-05 (Actual); Study Completion 2014-05-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Period I (443 participants) was a Pre-study screening period. Period II (186 participants) was a Run-in period in which participants received open-label montelukast (ML) 10 mg and matching single-blind placebo once daily (QD). Whereas 443 participants were screened, 107 eligible participants were enrolled and randomized to treatment in Period III.
Groups:
- MK-1029 + ML → Placebo + ML: Participants received 4 weeks of MK-1029 150 mg QD + ML 10 mg QD in Period III and Placebo + ML 10 mg QD in Period V. Period IV was a 4-week wash-out period during which participants received single-blind Placebo QD and open-label ML 10 mg QD.
- Placebo + ML → MK-1029 + ML: Participants received 4 weeks of Placebo QD + ML 10 mg QD in Period III and MK-1029 150 mg QD + ML 10 mg QD in Period V. Period IV was a 4-week wash-out period during which participants received single-blind Placebo QD and open-label ML 10 mg QD.
Period: Period III of Treatment (4 Weeks)
Arm/Group | MK-1029 + ML → Placebo + ML | Placebo + ML → MK-1029 + ML
Started | 54 | 53
Completed | 47 | 45
Not Completed | 7 | 8
Not completed — Lack of Efficacy | 0 | 2
Not completed — Non-Compliance with Protocol | 1 | 2
Not completed — Physician Decision | 5 | 3
Not completed — Protocol Violation | 1 | 0
Not completed — Adverse Event | 0 | 1
Period: Period IV Washout (4 Weeks)
Arm/Group | MK-1029 + ML → Placebo + ML | Placebo + ML → MK-1029 + ML
Started | 47 | 45
Completed | 44 | 42
Not Completed | 3 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 2 | 0
Not completed — Non-Compliance with Study Drug | 0 | 1
Period: Period V of Treatment (4 Weeks)
Arm/Group | MK-1029 + ML → Placebo + ML | Placebo + ML → MK-1029 + ML
Started | 44 | 42
Completed | 39 | 42
Not Completed | 5 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 3 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- MK-1029 150 mg + ML → Placebo + ML: Participants received 4 weeks of MK-1029 150 mg QD + ML 10 mg QD in Period III and Placebo + ML 10 mg QD in Period V. Period IV was a 4-week wash-out period during which participants received single-blind Placebo QD and open-label ML 10 mg QD
- Placebo + ML → MK-1029 150 mg + ML: Participants received 4 weeks of Placebo QD + ML 10 mg QD in Period III and MK-1029 150 mg QD + ML 10 mg QD in Period V. Period IV was a 4-week wash-out period during which participants received single-blind Placebo QD and open-label ML 10 mg QD
- Total: Total of all reporting groups
Arm/Group | MK-1029 150 mg + ML → Placebo + ML | Placebo + ML → MK-1029 150 mg + ML | Total
Number analyzed (Participants) | 54 | 53 | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (11.2) | 39.1 (13.5) | 40.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 38 | 73
  Male | 19 | 15 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 34 | 30 | 64
  Not Hispanic or Latino | 20 | 23 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 2 | 6
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 19 | 22 | 41
  More than one race | 29 | 28 | 57
  Unknown or Not Reported | 0 | 0 | 0
Forced Expiratory Volume in One Second (FEV1) [Mean (Standard Deviation); unit: Liters] — Population: Baseline was predose on the first day of treatment Period III
  Liters | 2.333 (0.637) | 2.243 (0.600) | 2.289 (0.618)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Forced Expiratory Volume in One Second (FEV1) at Week 4
Description: The change from baseline in FEV1 at Week 4 following treatment with MK-1029 + ML or placebo + ML was assessed. The pre-bronchodilator FEV1 was evaluated to assess the response to treatment for asthma. The primary efficacy evaluation period was the last week of each treatment period: Period III (Initial Therapy, Week 4) and Period V (Crossover Therapy, Week 4). The change from baseline in FEV1 was evaluated using a longitudinal data analysis (LDA) model with repeated measurements of FEV1, with treatment, visit, treatment-by-visit interaction, and period as fixed effects, and participant as random effect. Baseline FEV1 is defined as the measurement taken before dosing in each treatment period (i. e., at Visit 3 [Week 0], prior to Period III and at Visit 6 [Week 8], prior to Period V). The Baseline Characteristics section shows FEV1 values at baseline.
Time Frame: The week before the first dose in Period III or V (Baseline) and the last week of Period III or V
Population: All randomized participants who received at least one dose of study treatment in any crossover period (i.e., Period III or Period V), and had at least one measurement for the outcome analysis, as well as a pre-dose baseline measurement.
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- MK-1029 + ML: Participants received 4 weeks treatment with MK-1029 150 mg QD + ML 10 mg QD in Period III or V. Period IV was a 4-week washout period during which participants received single-blind Placebo QD and open-label ML 10 mg QD
- Placebo + ML: Participants received 4 weeks treatment with Placebo QD + ML 10 mg QD in Period III or V. Period IV was a 4-week wash-out period during which participants received single-blind Placebo QD and open-label ML 10 mg QD
Arm/Group | MK-1029 + ML | Placebo + ML
Number analyzed (Participants) | 93 | 97
Liters | 0.065 [0.003 to 0.126] | 0.017 [-0.044 to 0.078]
Statistical Analysis 1: Comparison: MK-1029 + ML vs Placebo + ML; Test type: Superiority; p = 0.282, LDA model; The LDA model assumes that repeated measurements follow a multivariate normal distribution; Difference in Least Squares (LS) Means = 0.047, 95% CI 2-sided [-0.039 to 0.134]

2. Primary Outcome: Adverse Events During Treatment and Follow-up
Description: The number of participants who had at least one adverse event (AE) during study treatment and follow-up was assessed. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product. The number of participants with at least one AE was assessed. The number of participants in any treatment group with at least one AE was assessed.
Time Frame: Up to 14 days after the last dose in Period III or Period V (up to 6 weeks)
Population: All randomized participants who received at least one dose of study treatment and had follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1029 + ML | Placebo + ML
Number analyzed (Participants) | 96 | 97
Participants | 30 | 33

3. Primary Outcome: Discontinuation of Treatment Due to An Adverse Event
Description: The number of participants who discontinued study treatment due to an AE was assessed. An AE is defined as any unfavorable and unintended change in the structure, function, or chemistry of the body temporally associated with the use of the SPONSOR's product, whether or not considered related to the use of the product.
Time Frame: Up to the last dose in Period III or Period V (up to 4 weeks)
Population: All randomized participants who received at least one dose of study treatment and had follow-up.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1029 + ML | Placebo + ML
Number analyzed (Participants) | 96 | 97
Participants | 2 | 2

4. Secondary Outcome: Change From Baseline in Daytime Symptom Score (DSS) at Week 4
Description: The change from baseline in DSS at Week 4 following treatment was assessed. Participants used an electronic diary (e-Diary) to enter their asthma symptom scores every evening. Participants scored daily symptoms (chest discomfort, wheezing, shortness of breath, and cough) by responding to 4 questions: 1) Symptom frequency (0 = None of the time, 6 = All of the time); 2) Bothersomeness (0 = Not bothered, 6 = Severely bothered); 3) Activity limitation (0 = Not limited, 6 = Totally limited); 4) Frequency of activity limitation (0 = None of the time, 6 = All of the time). The average of the 4 scores for overall DSS ranges from 0 to 6 where a higher average indicates greater symptom severity. The average overall DSS was calculated over the week-long assessment periods. The change from baseline in DSS was evaluated using the LDA model with repeated measurements of DSS, with treatment, visit, treatment-by-visit interaction, and period as fixed effects, and participant as random effect.
Time Frame: The week before the first dose in Period III or V (Baseline) and the last week of Period III or V
Population: All randomized participants who received at least one dose of study treatment in any crossover period (i.e., Period III or Period V), and had at least one measurement for the outcome analysis.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MK-1029 + ML | Placebo + ML
Number analyzed (Participants) | 91 | 97
Score on a scale
  Baseline | 1.93 (0.91) | 1.98 (0.90)
  Change from Baseline at Week 4 | -0.18 (0.73) | -0.08 (0.64)

5. Secondary Outcome: Change From Baseline in Short-Acting Beta Agonist (SABA) Use at Week 4
Description: The change from baseline in SABA use at Week 4 after treatment with MK-1029 + ML or placebo + ML was assessed. Participants used the e-Diary upon arising and before going to sleep to enter the total number of SABA puffs used for asthma relief. The number of SABA puffs recorded was the number of canister actuations (e. g., when SABA use was required and 3 puffs were inhaled, this was recorded as 3). Participants also recorded the number of nebulizer treatments (1 nebulized SABA use = 3 puffs). The average daily number of puffs for an individual participant was calculated over the week-long assessment periods. The change from baseline in SABA use was evaluated using the LDA model with repeated measurements of SABA use, with treatment, visit, treatment-by-visit interaction, and period as fixed effects, and participant as random effect.
Time Frame: The week before the first dose in Period III or V (Baseline) and the last week of Period III or V
Population: All randomized participants who received at least one dose of study treatment in any crossover period (i.e., Period III or Period V), and had at least one measurement for the outcome analysis. A participant in the Placebo + ML arm received treatment in both Period III and Period V, and resulted in 98 measurements from 97 participants.
Measure: Mean (Standard Deviation); unit: Number of puffs
Units Other Than Participants: SABA Use Measurements
Arm/Group | MK-1029 + ML | Placebo + ML
Number analyzed (Participants) | 94 | 97
Number analyzed (SABA Use Measurements) | 94 | 98
Number of puffs
  Baseline | 3.203 (2.502) | 3.597 (2.018)
  Change from Baseline at Week 4 | -0.595 (1.995) | -0.561 (1.768)

6. Secondary Outcome: Change From Baseline in Nocturnal Awakenings at Week 4
Description: The change from baseline in nocturnal awakenings due to asthma at Week 4 after treatment with MK-1029 + ML or placebo + ML was assessed. The participant scored nocturnal awakenings by answering the question, "Did you wake up with asthma symptoms in the middle of the night or upon awakening in the morning?" (No or Yes). Participants recorded in the e-Diary the number of nights per week in which they awakened with asthma, as determined by dividing the number of nights of awakening with asthma by the total number of nights and then multiplying by 7 (standardized to a 7-day period). The change from baseline in nocturnal awakenings was evaluated using the LDA model with repeated measurements of nocturnal awakenings, with treatment, visit, treatment-by-visit interaction, and period as fixed effects, and participant as random effect.
Time Frame: The week before the first dose in Period III or V (Baseline) and the last week of Period III or V
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Number of nocturnal awakenings
Arm/Group | MK-1029 + ML | Placebo + ML
Number analyzed (Participants) | 69 | 74
Number of nocturnal awakenings
  Baseline | 4.97 (2.60) | 4.90 (2.62)
  Change from Baseline at Week 4 | -1.13 (2.16) | -1.30 (2.29)

7. Secondary Outcome: Change From Baseline in Morning (AM) Peak Expiratory Flow (PEF) at Week 4
Description: The change from baseline in AM PEF at Week 4 after treatment with MK-1029 + ML or placebo + ML was assessed in 97 participants. Participants performed triplicate AM PEF measurements in the morning upon rising. Participants entered all 3 measurements and the greatest AM PEF value was recorded by the e-Diary. Participants refrained from SABA use within the 4 hours prior to performing PEF measurements. The average AM PEF for an individual participant was calculated over the week-long assessment periods. The change from baseline in AM PEF was evaluated using the LDA model with repeated measurements of AM PEF, with treatment, visit, treatment-by-visit interaction, and period as fixed effects, and participant as random effect.
Time Frame: The week before the first dose in Period III or V (Baseline) and the last week of Period III or V
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Liters/min
Units Other Than Participants: AM PEF Measurements
Arm/Group | MK-1029 + ML | Placebo + ML
Number analyzed (Participants) | 93 | 97
Number analyzed (AM PEF Measurements) | 93 | 98
Liters/min
  Baseline | 336.57 (117.02) | 333.07 (110.65)
  Change from Baseline at Week 4 | 7.14 (41.86) | -2.70 (32.33)

8. Secondary Outcome: Change From Baseline in Evening (PM) PEF at Week 4
Description: The change from baseline in PM PEF at Week 4 after treatment with MK-1029 + ML or placebo + ML was assessed. Participants performed triplicate PM PEF measurements in the evening, immediately before study drug administration, at bedtime. Participants entered all 3 measurements and the greatest PM PEF value was recorded by the e-Diary. Participants refrained from SABA use within the 4 hours prior to performing PEF measurements. The average PM PEF for an individual participant was calculated over the week-long assessment periods. The change from baseline in PM PEF was evaluated using the LDA model with repeated measurements of PM PEF, with treatment, visit, treatment-by-visit interaction, and period as fixed effects, and participant as random effect.
Time Frame: Baseline (Week 0 and Week 8), Last week of the 4-week treatment period
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters/min
Arm/Group | MK-1029 + ML | Placebo + ML
Number analyzed (Participants) | 91 | 96
Liters/min
  Baseline | 350.34 (121.45) | 342.30 (115.86)
  Change from Baseline at Week 4 | 8.25 (42.18) | -4.68 (34.47)

9. Secondary Outcome: Change From Baseline in Asthma Control Questionnaire (ACQ) Score at Week 4
Description: The change from baseline in the ACQ score at Week 4, after treatment, was assessed in 97 participants. Participants completed 6 items of the ACQ (i. e., ACQ-6) and provided the average of responses over the past week: 1) Frequency of nocturnal awakenings (0 = Never, 6 = Unable to sleep); 2) Symptom severity (0 = None, 6 = Very severe); 3) Activity limitations (0 = Not limited, 6 = Totally limited); 4) Breathlessness (0 = None, 6 = Very great deal); 5) Wheezing (0 = Not at all, 6 = All the time); 6) Daily SABA use (0 = None, 6 = More than 16 puffs on most days). The ACQ score ranges from 0 to 6 where a lower score indicates greater performance. The investigator reviewed the participant-completed ACQ-6 to ensure its completeness. The change from baseline in the ACQ score was evaluated using the LDA model with repeated measurements of the ACQ score, with treatment, visit, treatment-by-visit interaction, and period as fixed effects, and participant as random effect.
Time Frame: The week before the first dose in Period III or V (Baseline) and the last week of Period III or V
Population: All randomized participants who received at least one dose of study treatment in any crossover period (i.e., Period III or Period V), and had at least one measurement for the outcome analysis. A participant in the Placebo + ML arm received treatment in both Period III and Period V, and resulted in 99 measurements from 97 participants.
Measure: Mean (Standard Deviation); unit: Score on a scale
Units Other Than Participants: ACQ Measurements
Arm/Group | MK-1029 + ML | Placebo + ML
Number analyzed (Participants) | 97 | 97
Number analyzed (ACQ Measurements) | 97 | 99
Score on a scale
  Baseline | 2.09 (0.84) | 2.25 (0.86)
  Change from Baseline at Week 4 | -0.49 (0.86) | -0.48 (0.99)

ADVERSE EVENTS:
Time Frame: Up to 14 days after the last dose in Period III or Period V (up to 6 weeks)
Groups:
- MK 1029 + ML: Participants received 4 weeks treatment with MK-1029 150 mg QD + ML 10 mg QD in Period III or V. Period IV was a 4-week wash-out period during which participants received single-blind Placebo QD and open-label ML 10 mg QD.
Arm/Group | MK 1029 + ML | Placebo + ML
All-Cause Mortality (participants affected / at risk) | 0/96 | 0/97
Serious Adverse Events (participants affected / at risk) | 0/96 | 0/97
Other Adverse Events (participants affected / at risk) | 14/96 | 14/97
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK 1029 + ML (N=96) | Placebo + ML (N=97)
Nasopharyngitis (Infections and infestations) | 8 (9) | 8 (8)
Asthma (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This study is intended for publication, even if terminated prematurely. The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.